CLINICAL TRIAL: NCT01188148
Title: Series Studies of Bipolar Disorder-Valproate add-on Memantine Treatment
Brief Title: Series Studies of Bipolar Disorder-Valproate add-on Memantine
Acronym: MM
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: National Cheng-Kung University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BPMM HR-98-025
Record Dates: First submitted 2010-08-23; First posted 2010-08-25 (Estimated); Last update posted 2013-09-17 (Estimated); Status verified 2009-08

CONDITIONS: Bipolar Disorders
MeSH Terms: conditions — Bipolar Disorder | interventions — Memantine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- VPA & Placebo (Active Comparator): VPA & Placebo
  Interventions: Drug: Placebo
- VPA & memantine (Experimental)
  Interventions: Drug: Memantine

INTERVENTIONS:
Drug: Memantine — 5 mg per day of memantine
  Arms: VPA & memantine
Drug: Placebo
  Arms: VPA & Placebo

SUMMARY:
All participants should fulfill the following criteria: aged between 18 and 65 years old, and of domestic Han descendants. Participants will be randomly assigned to either the (1) pharmacotherapy (valproate add-on memantine) group; (2) pharmacotherapy (valproate add-on memantine) plus Cognitive Behavior Group Therapy (CBGT) group; (3) valproate add-on placebo plus CBGT group, or (4) valproate add-on placebo only group. A total of 240-320 individuals (60-80 participants per group) will be recruited for this study. For each CBGT group, 12-weekly sessions are scheduled according to patients' preference. The investigators will attempt to understand the effects of pharmaceutical drugs for mood stabilizers add-on neuro-protective drugs, pharmacotherapy with CBGT, mood stabilizer with CBGT, and the use of only traditional mood stabilizers in the treatment of BP II. Comparisons will be made for each type of treatment and possible mechanisms will be examined regarding the pharmacotherapy and CBGT for bipolar disorder patients.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patient aged >=18 and <= 65 years.
2. A diagnosis of bipolar II disorder according to DSM-IV-TR criteria made by a specialist in psychiatry.
3. A total of HDRS score at least 18 or YMRS score at least 14 at screen.
4. Signed informed consent by patient or legal representative.

Exclusion Criteria:

1. Women of childbearing potential not using adequate contraception as per investigator judgment or not willing to comply with contraception for duration of study.
2. Females who are pregnant or nursing.
3. Patient has received memantine or other selective cyclo-oxygenase 2 (Cox-2) inhibitors within 1 week prior to first dose of double-blind medication.
4. Axis-I DSM-IV-TR diagnosis other than bipolar II disorder.
5. Current evidence of an uncontrolled and/or clinically significant medical condition (e.g., cardiac, hepatic and renal failure), which in the judgments of the investigator, would compromise patient safety or preclude study participation.
6. History of intolerance to valproate or memantine or other Cox-2 inhibitors.
7. History of sensitivity reaction (e.g., urticaria, angioedema, bronchospasm, severe rhinitis, anaphylactic shock) precipitated by memantine
8. Patient has received electroconvulsive therapy (ECT) within 4 weeks prior to first dose of doubleblind medication.
9. Inclusion in another bipolar disorder study or study for another indication with psychotropic's within the last 30 days prior to start of study.
10. Increase in total SGOT, SGPT, BUN and creatinine by more than 3X ULN (upper limit of normal).
11. Substance-related disorders within 6 months prior to study start, borderline personality disorder, schizophrenia, or other major psychiatric disorders as defined by DSM-IV criteria.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 219 (Actual)
Dates: Start 2009-08; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Young's Mania Rating Scale (YMRS) | baseline, 1, 2, 4, 8 and 12 weeks
  Normally, YMRS is used to evaluate the Bipolar Disorder Patient's mood change.
Hamilton Depression Rating Scale (HDRS) | baseline, 1, 2, 4, 8 and 12 weeks
  Normally, YMRS is used to evaluate the Bipolar Disorder Patient's mood change of depression.

SECONDARY OUTCOMES:
cytokines | baseline, 1, 2, 4, 8 and 12 weeks
Clinical Global Impression (CGI) | baseline, 1, 2, 4, 8 and the week 12
  CGI will be used to evaluate how the patient's adverse effect go on during the trial.
lipid profiles | baseline, 1, 2, 4, 8 and 12 weeks
  HDL, LDL, cholesterol and etc.

OTHER OUTCOMES:
genetics | baseline
  ALDH2, ADH1B, COMT, DRD2, DRD3, BDNFVal66Met

CONTACTS AND LOCATIONS:
Overall Officials: Ru-Band Lu, MD, Principal Investigator — National Cheng-Kung University Hospital
Locations (1):
- Ru-Band Lu, Tainan, Taiwan

REFERENCES:
- [Derived] Lee SY, Chen SL, Chang YH, Chen SH, Chu CH, Huang SY, Tzeng NS, Wang CL, Wang LJ, Lee IH, Yeh TL, Yang YK, Hong JS, Lu RB. Genotype variant associated with add-on memantine in bipolar II disorder. Int J Neuropsychopharmacol. 2014 Feb;17(2):189-97. doi: 10.1017/S1461145713000825. Epub 2013 Oct 9. PMID 24103632
- [Derived] Lee SY, Chen SL, Chang YH, Chen PS, Huang SY, Tzeng NS, Wang YS, Wang LJ, Lee IH, Yeh TL, Yang YK, Lu RB, Hong JS. Add-on memantine to valproate treatment increased HDL-C in bipolar II disorder. J Psychiatr Res. 2013 Oct;47(10):1343-8. doi: 10.1016/j.jpsychires.2013.06.017. Epub 2013 Jul 18. PMID 23870798
- [Derived] Lee SY, Chen SL, Chang YH, Chen PS, Huang SY, Tzeng NS, Wang YS, Wang LJ, Lee IH, Wang TY, Yeh TL, Yang YK, Hong JS, Lu RB. Inflammation's Association with Metabolic Profiles before and after a Twelve-Week Clinical Trial in Drug-Naive Patients with Bipolar II Disorder. PLoS One. 2013 Jun 27;8(6):e66847. doi: 10.1371/journal.pone.0066847. Print 2013. PMID 23826157